CLINICAL TRIAL: NCT06272253
Title: Immunobridging Study: Immunogenicity and Safety of INAVAC (Vaksin Merah Putih - UNAIR SARS-CoV-2 (Vero Cell Inactivated)) as Heterologue Booster in Adolescent Subjects in Indonesia
Brief Title: UNAIR Inactivated COVID-19 Vaccine INAVAC as Heterologue Booster (Immunobridging Study) in Adolescent Subjects
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Dr. Soetomo General Hospital (Other Government)
Collaborators: Indonesia-MoH (Other Government); Universitas Airlangga (Other); PT Biotis Pharmaceuticals, Indonesia (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UNAIR-MP-INAKTIF-R-010
Record Dates: First submitted 2024-02-18; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: COVID-19 Pandemic; COVID-19 Vaccines
Keywords: Inactivated COVID-1 9 Vaccine; Immunobridging Study; Immunogenicity; Safety; COVID-19; Indonesia
MeSH Terms: conditions — COVID-19 | interventions — vaksin merah putih - UA SARS-CoV-2 COVID-19 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- INAVAC (Vaksin Merah Putih - UA-SARS CoV-2 (Vero Cell Inactivated) 5 μg (Experimental): Study product are provided in the form of liquid in vial single dose (0.5 ml). The vaccine will be given 1 dose (0.5 ml) once.
  Interventions: Biological: INAVAC (Vaksin Merah Putih - UA- SARS CoV-2 (Vero Cell Inactivated) 5 μg

INTERVENTIONS:
Biological: INAVAC (Vaksin Merah Putih - UA- SARS CoV-2 (Vero Cell Inactivated) 5 μg — Dose : 1 dose 0.5 ml containing 5 μg inactivated SARS-CoV-2 virus, Tween 80, histidine, Polysorbate 80, Aluminium hydroxide gel, and sodium chloride.

SUMMARY:
This is an open label trial. There will only be 1 group in the study. All subjects will receive INAVAC vaccine and be followed for 6 months.

The vaccine will be administered intramuscularly. This study will be started after the interim analysis of the phase III INAVAC trial in adolescent. This study will have two interim and one full analysis reports.

DETAILED DESCRIPTION:
This is an open label trial. There will only be 1 group in the study. All subjects will receive INAVAC vaccine and be followed for 6 months.

The vaccine will be administered intramuscularly. This study will be started after the interim analysis of the phase III INAVAC trial in adolescent. This study will have two interim and one full analysis reports.

Data Safety Monitoring Board will be commissioned for this study to evaluate safety data over the study period and to review any events that meet a specific study pausing rule or any other safety issue that may arise. They will review the 7 and 28 days safety data following the vaccine, and then the 3 and 6 months safety data. The immunogenicity data will be evaluated until 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females, adolescents age 12-17 years old. Healthy status will be determined by the investigator based on medical history, clinical laboratory results, vital sign measurements, and physical examination at screening.
2. Subjects already received 2 (two) doses of Coronavac (Sinovac) vaccines at least 3 months prior to this study.
3. Subjects and the parents or guardian have been informed properly regarding the study and signed the informed consent form
4. Subject and the parents or guardian will commit to comply with the instructions of the investigator and the schedule of the trial
5. Participants agree not to donate bone marrow, blood, and blood products from the first study vaccine administration until 3 months after receiving the vaccine.
6. Participants and the parents or guardian must be willing to provide verifiable identification, has means to be contacted and to contact the investigator during the study.

Exclusion Criteria:

1. Subjects concomitantly enrolled or scheduled to be enrolled in another vaccine trial
2. Evolving mild, moderate, and severe illness, especially infectious diseases or fever (axillary temperature 37.5oC or more) concurrent or within 7 days prior to study vaccination. This includes respiratory or constitutional symptms consistent with SARS-CoV-2 (cough, sore throat, difficulty in breathing, etc)
3. Known history of allergy to any component of the vaccines
4. History of uncontrolled coagulopathy or blood disorders contraindicating intramuscular injection
5. Any autoimmune or immunodeficiency disease/condition
6. Subjects who have received in the previous 4 weeks a treatment likely to alter the immune response (intravenous immunoglobulin, blood derived products, long term corticosteroid - more than 2 weeks, and so on), OR anticipation of the need for immunosuppressive treatment within 6 months after last vaccination. The use of topical or nasal steroid will be permitted. Inhaled glucocorticoids are prohibited.
7. Unstable chronic disease, inclusive of uncontrolled hypertension, congestive heart failure, chronic obstructive pulmonary disease, asthma, chronic urticaria, diabetes requiring use of medicine. The final decision regarding this condition will be decided by the attending field clinicians or investigator.
8. Any abnormality or chronic disease which according to the investigator might interfere with the assessment of the trial objectives
9. Subjects already immunized with any other vaccines within 4 weeks prior and expect to receive other vaccines within 60 days following the first dose
10. Individuals who have a previously ascertained Covid-19 in the period of 1 month (for mild, moderate, or asymptomatic people) or 3 months (for severe Covid-19) before the first recruit of this study, or in a close contact in the last 14 days with confirmed case of Covid-19.
11. Positive test for SARS-CoV-2 (Antigen or PCR) at screening prior to the vaccination. Testing may be repeated during the screening period if exposure to positive confirmed case of SARS-CoV-2 is suspected, at the discretion of investigator.
12. History of alcohol or substance abuse
13. HIV patients.
14. Malignancy patients within 3 years prior to study vaccination.
15. Any neurological disease or history of significant neurological disorder such as meningitis, encephalitis, Guillain-Barre Syndrome, multiple sclerosis, etc
16. Vital sign abnormalities and clinical laboratory abnormalities as decided by the investigators. Vital sign measurements and clinical laboratory testing may be repeated before the final decision.
17. Women who are pregnant or who plan to become pregnant during the study.
18. Participant has major psychiatric problem or illness
19. Participant cannot communicate reliably with the investigator
20. Participant has contraindication to intramuscular injection and blood draws, such as bleeding disorders or phobia.
21. Participant had major surgery within 12 weeks before vaccination which will not be fully recovered, or has major surgery planned during the time participant is expected to participate in the study or within 6 months after the vaccination.
22. Any condition that in the opinion of the investigators would pose a health risk to the subject if enrolled or could interfere with the evaluation of the vaccine or interpretation of the study results
23. Study team members.
24. Subject planning to move from the study area before the end of study period.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 250 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2024-03-19 (Estimated); Study Completion 2024-07-19 (Estimated)

PRIMARY OUTCOMES:
Humoral Immune Response (Neutralizing antibody) | 28 days after the booster vaccination
  SARS-CoV-2 Neutralization: SARS-CoV-2 neutralizing titers in serum measured by a virus neutralization assay, at 28 days following vaccination with INAVAC vaccine as heterologue booster in healthy adolescents age 12-17 years old.

SECONDARY OUTCOMES:
Incidence of Adverse Events | 7 and 28 days, 3 and 6 months following vaccination with INAVAC vaccine as heterologue booster.
  1. Solicited - clinical (local and systemic) adverse events for 7 and 28 days, 3 and 6 months following vaccination with INAVAC vaccine as heterologue booster administered intramuscularly in healthy adolescents age 12-17 years old.
  2. Unsolicited adverse events for 7 and 28 days, 3 and 6 months following vaccination with INAVAC vaccine as heterologue booster administered intramuscularly in healthy adolescents age 12-17 years old.
  3. Serious adverse events (SAE) throughout the study.
Humoral Immune Response - The neutralizing antibody | 3 and 6 months following vaccination with INAVAC vaccine as heterologue booster
  SARS-CoV-2 Neutralization: SARS-CoV-2 neutralizing titers in serum measured by a virus neutralization assay, for 3 and 6 months following vaccination with INAVAC vaccine as heterologue booster administered intramuscularly in healthy Adolescent subjects.
Humoral Immune Response-IgG SARS-CoV-2 neutralizing titer by CLIA | 28 days, 3 and 6 months following vaccination with INAVAC vaccine as heterologue booster
  IgG RBD SARS-CoV-2 (CLIA): analysis of IgG RBD SARS-CoV-2 antibodies for 3 and 6 months following vaccination with INAVAC vaccine as heterologue booster administered intramuscularly in healthy Adolescent subjects.

OTHER OUTCOMES:
Exploratory Endpoints-Whole Genome Sequencing | Through study completion, an average of 6 months after the study product administration
  Whole genome sequencing (WGS) of S protein of SARS-CoV-2 virus from positive Covid-19 cases

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Soetomo General Hospital, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang C, Wang Z, Wang G, Lau JY, Zhang K, Li W. COVID-19 in early 2021: current status and looking forward. Signal Transduct Target Ther. 2021 Mar 8;6(1):114. doi: 10.1038/s41392-021-00527-1. PMID 33686059
- [Result] Noh JY, Song JY, Yoon JG, Seong H, Cheong HJ, Kim WJ. Safe hospital preparedness in the era of COVID-19: The Swiss cheese model. Int J Infect Dis. 2020 Sep;98:294-296. doi: 10.1016/j.ijid.2020.06.094. Epub 2020 Jun 30. PMID 32619759
- [Result] Badan POM Republik Indonesia. Dowloaded from https://www.pom.go.id/new/ view/more/pers/605/Pastikan-Keamanan-danMutu-Vaksin---Badan-POM-Kawal- Uji-Klinik-Vaksin-Merah-Putih.html. Accessed 11 October 2021.
- [Result] Irwin A. What it will take to vaccinate the world against COVID-19. Nature. 2021 Apr;592(7853):176-178. doi: 10.1038/d41586-021-00727-3. No abstract available. PMID 33767468
- [Result] So AD, Woo J. Reserving coronavirus disease 2019 vaccines for global access: cross sectional analysis. BMJ. 2020 Dec 15;371:m4750. doi: 10.1136/bmj.m4750. PMID 33323376
- [Result] Biswas M, Rahaman S, Biswas TK, Haque Z, Ibrahim B. Association of Sex, Age, and Comorbidities with Mortality in COVID-19 Patients: A Systematic Review and Meta-Analysis. Intervirology. 2020 Dec 9:1-12. doi: 10.1159/000512592. Online ahead of print. PMID 33296901
- [Result] Polack FP, Thomas SJ, Kitchin N, Absalon J, Gurtman A, Lockhart S, Perez JL, Perez Marc G, Moreira ED, Zerbini C, Bailey R, Swanson KA, Roychoudhury S, Koury K, Li P, Kalina WV, Cooper D, Frenck RW Jr, Hammitt LL, Tureci O, Nell H, Schaefer A, Unal S, Tresnan DB, Mather S, Dormitzer PR, Sahin U, Jansen KU, Gruber WC; C4591001 Clinical Trial Group. Safety and Efficacy of the BNT162b2 mRNA Covid-19 Vaccine. N Engl J Med. 2020 Dec 31;383(27):2603-2615. doi: 10.1056/NEJMoa2034577. Epub 2020 Dec 10. PMID 33301246
- [Result] Baden LR, El Sahly HM, Essink B, Kotloff K, Frey S, Novak R, Diemert D, Spector SA, Rouphael N, Creech CB, McGettigan J, Khetan S, Segall N, Solis J, Brosz A, Fierro C, Schwartz H, Neuzil K, Corey L, Gilbert P, Janes H, Follmann D, Marovich M, Mascola J, Polakowski L, Ledgerwood J, Graham BS, Bennett H, Pajon R, Knightly C, Leav B, Deng W, Zhou H, Han S, Ivarsson M, Miller J, Zaks T; COVE Study Group. Efficacy and Safety of the mRNA-1273 SARS-CoV-2 Vaccine. N Engl J Med. 2021 Feb 4;384(5):403-416. doi: 10.1056/NEJMoa2035389. Epub 2020 Dec 30. PMID 33378609
- [Result] Voysey M, Clemens SAC, Madhi SA, Weckx LY, Folegatti PM, Aley PK, Angus B, Baillie VL, Barnabas SL, Bhorat QE, Bibi S, Briner C, Cicconi P, Collins AM, Colin-Jones R, Cutland CL, Darton TC, Dheda K, Duncan CJA, Emary KRW, Ewer KJ, Fairlie L, Faust SN, Feng S, Ferreira DM, Finn A, Goodman AL, Green CM, Green CA, Heath PT, Hill C, Hill H, Hirsch I, Hodgson SHC, Izu A, Jackson S, Jenkin D, Joe CCD, Kerridge S, Koen A, Kwatra G, Lazarus R, Lawrie AM, Lelliott A, Libri V, Lillie PJ, Mallory R, Mendes AVA, Milan EP, Minassian AM, McGregor A, Morrison H, Mujadidi YF, Nana A, O'Reilly PJ, Padayachee SD, Pittella A, Plested E, Pollock KM, Ramasamy MN, Rhead S, Schwarzbold AV, Singh N, Smith A, Song R, Snape MD, Sprinz E, Sutherland RK, Tarrant R, Thomson EC, Torok ME, Toshner M, Turner DPJ, Vekemans J, Villafana TL, Watson MEE, Williams CJ, Douglas AD, Hill AVS, Lambe T, Gilbert SC, Pollard AJ; Oxford COVID Vaccine Trial Group. Safety and efficacy of the ChAdOx1 nCoV-19 vaccine (AZD1222) against SARS-CoV-2: an interim analysis of four randomised controlled trials in Brazil, South Africa, and the UK. Lancet. 2021 Jan 9;397(10269):99-111. doi: 10.1016/S0140-6736(20)32661-1. Epub 2020 Dec 8. PMID 33306989
- [Result] Palacios R, Patino EG, de Oliveira Piorelli R, Conde MTRP, Batista AP, Zeng G, Xin Q, Kallas EG, Flores J, Ockenhouse CF, Gast C. Double-Blind, Randomized, Placebo-Controlled Phase III Clinical Trial to Evaluate the Efficacy and Safety of treating Healthcare Professionals with the Adsorbed COVID-19 (Inactivated) Vaccine Manufactured by Sinovac - PROFISCOV: A structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Oct 15;21(1):853. doi: 10.1186/s13063-020-04775-4. PMID 33059771
- [Result] Tanriover MD, Doganay HL, Akova M, Guner HR, Azap A, Akhan S, Kose S, Erdinc FS, Akalin EH, Tabak OF, Pullukcu H, Batum O, Simsek Yavuz S, Turhan O, Yildirmak MT, Koksal I, Tasova Y, Korten V, Yilmaz G, Celen MK, Altin S, Celik I, Bayindir Y, Karaoglan I, Yilmaz A, Ozkul A, Gur H, Unal S; CoronaVac Study Group. Efficacy and safety of an inactivated whole-virion SARS-CoV-2 vaccine (CoronaVac): interim results of a double-blind, randomised, placebo-controlled, phase 3 trial in Turkey. Lancet. 2021 Jul 17;398(10296):213-222. doi: 10.1016/S0140-6736(21)01429-X. Epub 2021 Jul 8. PMID 34246358
- [Result] Al Kaabi N, Zhang Y, Xia S, Yang Y, Al Qahtani MM, Abdulrazzaq N, Al Nusair M, Hassany M, Jawad JS, Abdalla J, Hussein SE, Al Mazrouei SK, Al Karam M, Li X, Yang X, Wang W, Lai B, Chen W, Huang S, Wang Q, Yang T, Liu Y, Ma R, Hussain ZM, Khan T, Saifuddin Fasihuddin M, You W, Xie Z, Zhao Y, Jiang Z, Zhao G, Zhang Y, Mahmoud S, ElTantawy I, Xiao P, Koshy A, Zaher WA, Wang H, Duan K, Pan A, Yang X. Effect of 2 Inactivated SARS-CoV-2 Vaccines on Symptomatic COVID-19 Infection in Adults: A Randomized Clinical Trial. JAMA. 2021 Jul 6;326(1):35-45. doi: 10.1001/jama.2021.8565. PMID 34037666
- [Result] Kyriakidis NC, Lopez-Cortes A, Gonzalez EV, Grimaldos AB, Prado EO. SARS-CoV-2 vaccines strategies: a comprehensive review of phase 3 candidates. NPJ Vaccines. 2021 Feb 22;6(1):28. doi: 10.1038/s41541-021-00292-w. PMID 33619260
- [Result] Mendonca SA, Lorincz R, Boucher P, Curiel DT. Adenoviral vector vaccine platforms in the SARS-CoV-2 pandemic. NPJ Vaccines. 2021 Aug 5;6(1):97. doi: 10.1038/s41541-021-00356-x. PMID 34354082
- [Result] Yadav T, Srivastava N, Mishra G, Dhama K, Kumar S, Puri B, Saxena SK. Recombinant vaccines for COVID-19. Hum Vaccin Immunother. 2020 Dec 1;16(12):2905-2912. doi: 10.1080/21645515.2020.1820808. Epub 2020 Nov 24. PMID 33232211
- [Result] Pollard AJ, Bijker EM. A guide to vaccinology: from basic principles to new developments. Nat Rev Immunol. 2021 Feb;21(2):83-100. doi: 10.1038/s41577-020-00479-7. Epub 2020 Dec 22. PMID 33353987
- [Result] Excler JL, Saville M, Berkley S, Kim JH. Vaccine development for emerging infectious diseases. Nat Med. 2021 Apr;27(4):591-600. doi: 10.1038/s41591-021-01301-0. Epub 2021 Apr 12. PMID 33846611
- [Result] Bhattacharya S, Dasgupta R. Smallpox and polio eradication in India: comparative histories and lessons for contemporary policy. Cien Saude Colet. 2011 Feb;16(2):433-44. doi: 10.1590/s1413-81232011000200007. PMID 21340319
- [Result] Jayk Bernal A, Gomes da Silva MM, Musungaie DB, Kovalchuk E, Gonzalez A, Delos Reyes V, Martin-Quiros A, Caraco Y, Williams-Diaz A, Brown ML, Du J, Pedley A, Assaid C, Strizki J, Grobler JA, Shamsuddin HH, Tipping R, Wan H, Paschke A, Butterton JR, Johnson MG, De Anda C; MOVe-OUT Study Group. Molnupiravir for Oral Treatment of Covid-19 in Nonhospitalized Patients. N Engl J Med. 2022 Feb 10;386(6):509-520. doi: 10.1056/NEJMoa2116044. Epub 2021 Dec 16. PMID 34914868
- [Result] Mahase E. Covid-19: Pfizer's paxlovid is 89% effective in patients at risk of serious illness, company reports. BMJ. 2021 Nov 8;375:n2713. doi: 10.1136/bmj.n2713. No abstract available. PMID 34750163
- [Result] Abbasi J. Studies Suggest COVID-19 Vaccine Boosters Save Lives. JAMA. 2022 Jan 11;327(2):115. doi: 10.1001/jama.2021.23455. No abstract available. PMID 35015054
- [Result] Burckhardt RM, Dennehy JJ, Poon LLM, Saif LJ, Enquist LW. Are COVID-19 Vaccine Boosters Needed? The Science behind Boosters. J Virol. 2022 Feb 9;96(3):e0197321. doi: 10.1128/JVI.01973-21. Epub 2021 Nov 24. PMID 34817198
- [Result] Mattiuzzi C, Lippi G. Efficacy of COVID-19 vaccine booster doses in older people. Eur Geriatr Med. 2022 Feb;13(1):275-278. doi: 10.1007/s41999-022-00615-7. Epub 2022 Jan 24. PMID 35067909
- [Result] Parker EPK, Desai S, Marti M, Nohynek H, Kaslow DC, Kochhar S, O'Brien KL, Hombach J, Wilder-Smith A. Response to additional COVID-19 vaccine doses in people who are immunocompromised: a rapid review. Lancet Glob Health. 2022 Mar;10(3):e326-e328. doi: 10.1016/S2214-109X(21)00593-3. No abstract available. PMID 35180408
- See also: New York Vaccine Tracker. Downloaded from https://www.nytimes.com/interactive/2020/science/coronavirus-vaccine- tracker.html. Accessed 30 April 2022. — https://www.nytimes.com/interactive/2020/science/coronavirus-vaccine-tracker.html
- See also: Badan POM Republik Indonesia. Dowloaded from https://www.pom.go.id/siaran-pers/pastikan-keamanan-dan-mutu-vaksin-badan-pom-kawal-uji-klinik-vaksin-merah-putih. Accessed 11 October 2021. — https://www.pom.go.id/siaran-pers/pastikan-keamanan-dan-mutu-vaksin-badan-pom-kawal-uji-klinik-vaksin-merah-putih
- See also: Worldometer coronavirus cases. Downloaded from https://www.worldometers.info/coronavirus/. Accessed 30 April 2022. — https://www.worldometers.info/coronavirus/